CLINICAL TRIAL: NCT06808282
Title: Effects of Dark Chocolate on the Risk Factors of Cardiovascular Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 658065
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White chocolate (Active Comparator): Subjects consume 50g of white chocolate daily for 15 days.
  Interventions: Other: White chocolate
- Dark chocolate (Experimental): Subjects consume 50g of dark chocolate daily for 15 days.
  Interventions: Other: Dark chocolate

INTERVENTIONS:
Other: White chocolate — To determine the effects of white chocolate consumption on risk factors of cardiovascular diseases
  Arms: White chocolate
Other: Dark chocolate — To determine the effects of dark chocolate consumption on risk factors of cardiovascular diseases
  Arms: Dark chocolate

SUMMARY:
Cardiovascular disease (CVD) is the number one cause of death in the US. Epidemiologic evidence supports that antioxidant-rich diets promote health and attenuate or delay the onset of CVD. Cocoa and chocolate products have among the highest antioxidant concentrations compared to other antioxidant food sources. The objective of this study is to examine the effects of regular dark chocolate, bloomed dark chocolate, and white chocolate on cardiovascular health markers.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects

Exclusion Criteria:

* Smoker
* Pregnant woman
* Lactose intolerance
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to cacao

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of systolic and diastolic blood pressure | Baseline and Day 15
  Change of systolic and diastolic blood pressure will be determined to examine effects of dark chocolate consumption vs white chocolate.
Change of skin blood flow level | Baseline and Day 15
  Change of skin blood flow level will be determined using Laser Doppler Flowmetry to examine effects of dark chocolate consumption vs white chocolate. Laser Doppler flowmetry is an optical technology widely used in research to measure blood flow. It is a non-invasive, painless technique for studying microcirculatory changes in tissue.
Change of HDL cholesterol level | Baseline and Day 15
  Change of blood cholesterol level will be determined to examine effects of dark chocolate consumption vs white chocolate.
Change of antioxidant levels | Baseline and Day 15
  Change of antioxidant levels will be determined to examine effects of dark chocolate consumption vs white chocolate.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data collected in this study are used exclusively within the primary research group and will not be shared with other external researchers.